CLINICAL TRIAL: NCT00146705
Title: Long Term Follow-up of Pegylated-Interferon Alpha-2b and Lamivudine Combination Therapy in Patients With Chronic HBV Infection
Brief Title: Long Term Follow-up of Pegylated-Interferon Alpha-2b
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Other Study IDs: LTFU HBV 99-01
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Hepatitis B
Keywords: chronic HBV; Peginterferon; long term follow-up
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood samples are taken once

SUMMARY:
The aim of this study was to investigate the long term outcome of Peginterferon alpha-2b with or without the addition of lamivudine in patients with chronic hepatitis B

DETAILED DESCRIPTION:
Interferon alpha therapy is a generally accepted agent for the treatment of chronic HBV infection and effective in about one third of patients. Recently, in the HBV 99-01 study, pegylated interferon alpha-2b (PEG-IFN) has been shown to be effective in HBeAg-positive patients with chronic hepatitis B. In this study, 266 patients were randomized to receive PEG-IFN in combination with either lamivudine or placebo for 52 weeks.

Thirty-six percent of patients receiving monotherapy and thirty-five percent receiving combination therapy had lost serum HBeAg at the end of the 26 week post-treatment follow-up period and there was no difference between treatment groups (P = 0.91). More patients on combination therapy initially seroconverted (44% of patients, compared with 29% on monotherapy; P = 0.01) at the end of treatment but relapsed during follow-up. Similar response patterns were seen when response was assessed by DNA suppression and change in ALT levels.

In contrast to nucleoside analogues, such as lamivudine and adefovir dipivoxil, the virological and biochemical response to standard alpha-interferon has been shown to be durable after treatment discontinuation.In addition, standard alpha-interferon leads to improved survival and reduction of hepatocellular carcinoma in chronic hepatitis B patients.Pegylated interferons have shown to be effective in HBeAg-positive chronic hepatitis B patients, but the durability of the response and long-term outcome of treatment have yet to be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic Hepatitis B who participated in the HBV 99-01 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2005-05; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD PhD, Principal Investigator — Department of Gastroenterology and Hepatology, University Medical Center Rotterdam, Rotterdam, the Netherlands
Locations (1):
- University Medical Center Rotterdam, Rotterdam, Dr Molewaterplein 40, Netherlands

REFERENCES:
- [Background] Janssen HL, van Zonneveld M, Senturk H, Zeuzem S, Akarca US, Cakaloglu Y, Simon C, So TM, Gerken G, de Man RA, Niesters HG, Zondervan P, Hansen B, Schalm SW; HBV 99-01 Study Group; Rotterdam Foundation for Liver Research. Pegylated interferon alfa-2b alone or in combination with lamivudine for HBeAg-positive chronic hepatitis B: a randomised trial. Lancet. 2005 Jan 8-14;365(9454):123-9. doi: 10.1016/S0140-6736(05)17701-0. PMID 15639293
- [Background] van Zonneveld M, Honkoop P, Hansen BE, Niesters HG, Darwish Murad S, de Man RA, Schalm SW, Janssen HL. Long-term follow-up of alpha-interferon treatment of patients with chronic hepatitis B. Hepatology. 2004 Mar;39(3):804-10. doi: 10.1002/hep.20128. PMID 14999700
- [Background] van Nunen AB, Hansen BE, Suh DJ, Lohr HF, Chemello L, Fontaine H, Heathcote J, Song BC, Janssen HL, de Man RA, Schalm SW. Durability of HBeAg seroconversion following antiviral therapy for chronic hepatitis B: relation to type of therapy and pretreatment serum hepatitis B virus DNA and alanine aminotransferase. Gut. 2003 Mar;52(3):420-4. doi: 10.1136/gut.52.3.420. PMID 12584227
- [Derived] Brakenhoff SM, de Knegt RJ, van Campenhout MJH, van der Eijk AA, Brouwer WP, van Bommel F, Boonstra A, Hansen BE, Berg T, Janssen HLA, de Man RA, Sonneveld MJ. End-of-treatment HBsAg, HBcrAg and HBV RNA predict the risk of off-treatment ALT flares in chronic hepatitis B patients. J Microbiol Immunol Infect. 2023 Feb;56(1):31-39. doi: 10.1016/j.jmii.2022.06.002. Epub 2022 Jul 2. PMID 35941076
- [Derived] Brakenhoff SM, de Knegt RJ, Oliveira J, van der Eijk AA, van Vuuren AJ, Hansen BE, Janssen HLA, de Man RA, Boonstra A, Sonneveld MJ. Levels of Antibodies to Hepatitis B Core Antigen Are Associated With Liver Inflammation and Response to Peginterferon in Patients With Chronic Hepatitis B. J Infect Dis. 2022 Dec 28;227(1):113-122. doi: 10.1093/infdis/jiac210. PMID 35599306
- [Derived] Brakenhoff SM, de Man RA, Boonstra A, van Campenhout MJH, de Knegt RJ, van Bommel F, van der Eijk AA, Berg T, Hansen BE, Janssen HLA, Sonneveld MJ. Hepatitis B virus RNA decline without concomitant viral antigen decrease is associated with a low probability of sustained response and hepatitis B surface antigen loss. Aliment Pharmacol Ther. 2021 Jan;53(2):314-320. doi: 10.1111/apt.16172. Epub 2020 Nov 21. PMID 33222190
- [Derived] Buster EH, Flink HJ, Simsek H, Heathcote EJ, Sharmila S, Kitis GE, Gerken G, Buti M, de Vries RA, Verhey E, Hansen BE, Janssen HL. Early HBeAg loss during peginterferon alpha-2b therapy predicts HBsAg loss: results of a long-term follow-up study in chronic hepatitis B patients. Am J Gastroenterol. 2009 Oct;104(10):2449-57. doi: 10.1038/ajg.2009.371. Epub 2009 Jul 7. PMID 19584831